CLINICAL TRIAL: NCT06674681
Title: HPV Self-Collection Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HCI169477
Record Dates: First submitted 2024-10-29; First posted 2024-11-05 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-01

CONDITIONS: HPV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Self-Collection (Other): Patients at partnering clinics who are enrolled in the clinics' HPV self-collection program(s). The requirements for being enrolled in the program are based off of the American Cancer Society's recommendation for cervical cancer screening.
  Interventions: Diagnostic Test: HPV Self-Collection

INTERVENTIONS:
Diagnostic Test: HPV Self-Collection — HPV self-collection program for in-clinic and mailed cervical cancer screening.

SUMMARY:
The objective of the study is to develop, pilot, and analyze the effectiveness of HPV self-collection programs which will be used to follow up among women overdue for cervical cancer screening. The investigators will develop protocols for in-clinic and home-based HPV-self-collection programs and follow-up system for HPV-positive tests for community health centers and/or clinics. The program is meant to mail HPV-self-collection kits to women who are due and/or overdue for cervical cancer screening and the program is also meant to present women seen in clinic with a self-collection option for screening alongside a Pap test option. The research team will develop related informational resources on how to complete the test as well as information on screening options.

The study will neither experiment nor test the effectiveness of the self-collection process nor the assay of specimens for HPV and high-risk HPV strains. It is not a clinical investigation to assess the safety or effectiveness of a medical device. The study is implementation science and seeks to find optimal ways to implement this World Health Organization recommended screening option.

DETAILED DESCRIPTION:
There are 2 parts of this project; (i) the implementation of a self-collection program at clinics/FQHCs (which is a quality improvement project) and (ii) the study/research portion (which is implementation science).

(i) The investigators will develop protocols and educational materials for an HPV-self-collection program that is conducted in a healthcare setting and/or in patients' homes. These materials will inform individuals about HPV, cervical cancer, and other HPV-related cancers. They will also instruct individuals how to use a self-collection kit. The research team will adapt existing clinical protocol implementation documents for self-collection programs (e.g., colorectal screening, HIV screening, etc.) from available resources and our previous work and collaborations. Implementation protocol and workflows will be created to meet the needs of the individual clinics, and designed for adaptability for other clinics and scalability to other additional and larger health systems.

Self-collection Implementation. Our clinic partners will implement new protocols for cervical cancer screening and follow-up for positive screening results, as developed in earlier stages of the study and as quality improvement. A new option for screening-self-collection-will be offered to eligible patients as an in-clinic option (e.g., collection in the exam room, restroom, mobile clinic) as well as an at-home option. These options will be offered alongside (or after) a recommendation for the patient to receive a Pap test (a.k.a., Pap smear). Patients who test positive for HPV will be followed up with by the clinics to schedule an appointment where they can discuss the next steps with their healthcare provider.

This research will not test the effectiveness of the tools or assay on detecting HPV. Clinics plan for participants to use the Copan swab to self-collect a sample and this will be a dry collection; the specimen will not need to be suspended in a medium or other substance. Clinics will send specimens to an external laboratory that has already validated the assay of self-collected specimens with the Copan swab. The lab's procedures are consistent with regulations for lab developed tests (LDTs). Considering recent FDA approval for a couple of devices used for self-collection in the healthcare setting, clinics may adopt these approved devices for the current study.

Medical records review will not currently be done for research purposes, only for recruitment and/or reviewing study eligibility.

(ii) The investigators will identify and assess the current patient-level barriers and facilitators to HPV self-collection and/or regular, in-clinic HPV screening. Staff at our partner clinics will review their records to identify eligible patients. They will share a de-identified data set (with the exception of the patients' residential zip code, county, date of clinic visits, and medical record number) with our research team. The research team will use the zip codes and county information to code each patient's rurality status and other area-based measures. After coding for rurality, the research team will remove and/or destroy zip codes from our data set(s). Each participant will receive a unique identifier and our team will only store medical record numbers and clinic visit dates in a separate file with a link to the unique identifiers. This study will store this file on a server with security protocols the University deems acceptable for PHI. The file will be accessed by the minimum study personnel necessary.

Additionally, the research team will survey patients who participate in the program at 2 points to assess patient-level barriers to HPV self-collection and understand confusion, ease, and fidelity of both the self-collection process and instructions. Patients will be recruited as described in the recruitment section of this application. Participants will be consented using a questionnaire cover letter, a consenting process for which the researchers request documentation of consent be waived. The research team will collect respondents' names in order to link their data across the 2 surveys. At a future point, this study will seek approval for a medical records review during which the investigators will link some information from their medical records to these survey data.

After its implementation, this research will (1) survey healthcare team members; (2) interview healthcare team members; (3) conduct a records review of patient-level data to assess screening choices, completion, results, and follow up; and (4) conduct analysis of the workflow to evaluate the effectiveness of the self-collection protocol. The research team will evaluate the HPV self-collection program at the clinic- and organization-levels for program effectiveness, reach, barriers and facilitators to adoption, implementation, and maintenance. Finally, the research team will conduct a data synthesis to capitalize on the richness of the mixed methods approach.

ELIGIBILITY:
Inclusion Criteria:

* Women and individuals with a cervix.
* Aged 25-65 years during the study measurement period.
* Qualifying visit to the participating clinic.
* Overdue for cervical cancer screening.
* Those aged 24-64 who have not had cervical cytology (i.e., Pap test) performed within the last three and a half (3.5) years, or those aged 30-65 who have not had cervical HPV testing (i.e., primary HPV testing or contesting for HPV with Pap test) performed within the last five and a half (5.5) years.

Exclusion Criteria:

* Individuals without a cervix.
* Receiving hospice and/or palliative care during any part of the measurement period.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Clinic Level Implementation Rate | 1 year
  The proportion of people with a cervix who complete the test out of the number of people we were approached.

SECONDARY OUTCOMES:
At home utilization rate | 1 year
  The number of people who completed the test at home compared to the number of people who completed the test in clinic.
Follow-up care rate | 1 year
  Among those with positive HVP test results, the number of people who complete recommended care.

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Kepka, PhD, MPH, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Hospitals/Huntsman Cancer Institute Population Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No